CLINICAL TRIAL: NCT02611947
Title: CT Indexes of Emphysema and Airways in Healthy Volunteers: Normal Values; Relations With Gender, Height and Weight
Status: Completed | Type: Observational
Sponsor: Erasme University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: P2010/175
Record Dates: First submitted 2015-10-30; First posted 2015-11-23 (Estimated); Last update posted 2015-11-23 (Estimated); Status verified 2015-11

CONDITIONS: Healthy
Keywords: emphysema; airway remodelling; multidetector computed tomography
MeSH Terms: conditions — Emphysema; Airway Remodeling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Healthy Volunteers: Inclusion criteria:
  1. Aged 18 or more.
  2. Never smoked.
  3. No respiratory infection in the 4 weeks before the begin of the study.
  4. No history of pulmonary resection.
  5. No active malignancy or malignancy of any organ system within the past 5 years.
  Interventions: Radiation: Low-dose chest CT scans

INTERVENTIONS:
Radiation: Low-dose chest CT scans — Supine chest CT scan after full inspiration. Acquisition parameters: (Topogram 35 mA 120 kV 512 mm length)
  35 quality ref mAs with care-dose ON 120 kV Pitch 1.4 Rotation time 0.33 s Acquired images 64 x 0.6 mm

SUMMARY:
Various indexes have been proposed to quantify both pulmonary emphysema and airways disease on chest CT scans. It is unknown whether these indexes should be consider in absolute values or as compared to predicted normal values. The purposes of the present study is thus : a) to measure these indexes at CT in healthy volunteers; b) to investigate their relations with gender, height and weight.

DETAILED DESCRIPTION:
87 healthy volunteers performed consecutively a low-dose chest CT scan and pulmonary function tests:

1. On chest CT scans, indexes reflecting pulmonary emphysema and airways measurements have been computed by using dedicated softwares. Each of our three readers performed two reading sessions.

   Relative area of lung parenchyma with attenuation value less than -960 Hounsfield Units; luminal area and wall thickness in third and fourth generations airways were recorded.
2. Pulmonary function tests were performed: vital capacity, forced vital capacity , functional residual capacity, total lung capacity, residual volume, forced expiratory volume in one second, and diffusion lung capacity for carbon monoxide were recorded (either in absolute values and percentage of predicted values).

CT indexes were compared with gender, height and weight.

ELIGIBILITY:
Inclusion Criteria:

* Never smoked.
* No respiratory infection in the 4 weeks before the begin of the study.
* No history of pulmonary resection.
* No active malignancy or malignancy of any organ system within the past 5 years.

Exclusion Criteria:

* no exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy Volunteers
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2010-10; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
CT index - RA960 (%) | 4 hours
  From acquired data, images were reconstructed using a soft algorithm. On these soft images, the relative area of lung parenchyma with attenuation value less than -960 Hounsfield Units was computed (expressed in %), as an index representative of pulmonary emphysema extent.
CT index - LA3rd (mm2) | 4 hours
  From acquired data, images were reconstructed using a high resolution algorithm. On these high-resolution images, the airway lumen was measured in third generations of airways (expressed in mm2).
CT index - LA4th (mm2) | 4 hours
  From acquired data, images were reconstructed using a high resolution algorithm. On these high-resolution images, the airway lumen was measured in fourth generations of airways (expressed in mm2).
CT index - WT3rd (mm) | 4 hours
  From acquired data, images were reconstructed using a high resolution algorithm. On these high-resolution images, the airway wall was measured in third generations of airways (expressed in mm).
CT index - WT4th (mm) | 4 hours
  From acquired data, images were reconstructed using a high resolution algorithm. On these high-resolution images, the airway wall was measured in fourth generations of airways (expressed in mm).

SECONDARY OUTCOMES:
Pulmonary function tests - VC (l) | 4 hours
  Vital capacity was measured (expressed in l).
Pulmonary function tests - FVC (l) | 4 hours
  Forced vital capacity was measured (expressed in l).
Pulmonary function tests - FRC (l) | 4 hours
  Functional residual capacity capacity was measured (expressed in l).
Pulmonary function tests - TLC (l) | 4 hours
  Total lung capacity was measured (expressed in l).
Pulmonary function tests - RV (l) | 4 hours
  Residual volume was measured (expressed in l).
Pulmonary function tests - FEV1 (l) | 4 hours
  Forced expiratory volume in one second was measured (expressed in l).
Pulmonary function tests - DLCO (ml/min/ mmHg) | 4 hours
  Diffusion lung capacity for carbon monoxide was measured (expressed in ml/min/ mmHg)

CONTACTS AND LOCATIONS:
Overall Officials: Pierre Alain GEVENOIS, MD, PhD, Study Director — Erasme University Hospital
Locations (1):
- Erasme University Hospital, Brussels, Brussels Capital, Belgium

REFERENCES:
- [Background] Madani A, Zanen J, de Maertelaer V, Gevenois PA. Pulmonary emphysema: objective quantification at multi-detector row CT--comparison with macroscopic and microscopic morphometry. Radiology. 2006 Mar;238(3):1036-43. doi: 10.1148/radiol.2382042196. Epub 2006 Jan 19. PMID 16424242
- [Background] Madani A, De Maertelaer V, Zanen J, Gevenois PA. Pulmonary emphysema: radiation dose and section thickness at multidetector CT quantification--comparison with macroscopic and microscopic morphometry. Radiology. 2007 Apr;243(1):250-7. doi: 10.1148/radiol.2431060194. PMID 17392257
- [Background] Hackx M, Bankier AA, Gevenois PA. Chronic obstructive pulmonary disease: CT quantification of airways disease. Radiology. 2012 Oct;265(1):34-48. doi: 10.1148/radiol.12111270. PMID 22993219
- [Background] Hackx M, Gyssels E, Severo Garcia T, De Meulder I, Alard S, Bruyneel M, Van Muylem A, Ninane V, Gevenois PA. Chronic Obstructive Pulmonary Disease: CT Quantification of Airway Dimensions, Numbers of Airways to Measure, and Effect of Bronchodilation. Radiology. 2015 Dec;277(3):853-62. doi: 10.1148/radiol.2015140949. Epub 2015 May 19. PMID 25989594